CLINICAL TRIAL: NCT01136252
Title: Open-label Clinical Trial to Evaluate Safety and Efficacy of Intravitreal Adalimumab in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration Non-responders to the Conventional Treatment With Ranibizumab
Brief Title: Intravitreal Adalimumab in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZAPA-01/EudraCT 2009-017429-21; 2009-017429-21 (EudraCT Number)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Intravitreal adalimumab injection (0,1 ml= 50 mcg) in the eye of the included patients. Patients will be followed up every week for a total of 4 weeks, and after every month until 6 months. If it is necessary, repeat the injection every month, maximum three months
  Other Names: Humira®

SUMMARY:
Adalimumab is a humanized recombinant monoclonal antibody fragment targeted against tumor necrosis factor. This study will assess the safety and efficacy of intravitreal adalimumab administered in patients with choroidal neovascularization secondary to age-related macular degeneration non-responders to the conventional treatment with intravitreal ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

- Choroidal neovascularization secondary to age-related macular degeneration non-responders to the conventional treatment with ranibizumab (active choroidal neovascularization after loading phase of one injection per month for three consecutive months, followed by a maintenance phase with 5 injections in the last 12 months or 3 injections in the last 6 months

Exclusion Criteria:

* Only one functional eye
* Hypersensitivity to adalimumab or any component of the formulation
* Previous systemic treatment with adalimumab
* Cancer
* Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Patients proportion with electroretinogram alterations | 6 months

SECONDARY OUTCOMES:
Changes in retinal thickness measured by ocular coherence tomography | once a month to 6 months
Changes in best corrected visual acuity | once a month to 6 months
Incidence of adverse events | until 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Zapata, MD, Study Chair — Hospital Vall d'Hebron
Locations (1):
- Servicio de Oftalmologia. Hospital Universitario Vall d'Hebron, Barcelona, Barcelona, Spain